CLINICAL TRIAL: NCT05574764
Title: ABC Mental Health: A Behavioral Study of K-12 Teachers and School Staff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRO00111936; OT2HD107559 (NIH)
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Mental Health Wellness 1; Burnout, Professional; Self Efficacy
MeSH Terms: conditions — Burnout, Professional | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Teachers (Active Comparator): This cohort includes K-12 teachers. Schools will offer all teachers the professional development program called Cultivating Awareness and Resilience in Education (CARE) . CARE will be presented in three in-person training sessions over two to three months during the school year. Tools include mindful awareness practices and caring and emotion skills training. Each intervention workshop includes 30 to 35 participants and a facilitator, who is part of the CARE team. The workshops will be held at a location selected by the school, likely on their campus.
  Interventions: Behavioral: Cultivating Awareness and Resilience in Education (CARE)
- Staff, Non-Administrative (Active Comparator): This cohort includes non-administrative staff. Schools will offer all non-administrative staff the professional development program called Cultivating Awareness and Resilience in Education (CARE) . CARE will be presented in three in-person training sessions over two to three months during the school year. Tools include mindful awareness practices and caring and emotion skills training. Each intervention workshop includes 30 to 35 participants and a facilitator, who is part of the CARE team. The workshops will be held at a location selected by the school, likely on their campus.
  Interventions: Behavioral: Cultivating Awareness and Resilience in Education (CARE)
- Staff, Administrative (Active Comparator): This cohort includes administrative staff. Schools will offer all administrative staff the professional development program called Cultivating Awareness and Resilience in Education (CARE) . CARE will be presented in three in-person training sessions over two to three months during the school year. Tools include mindful awareness practices and caring and emotion skills training. Each intervention workshop includes 30 to 35 participants and a facilitator, who is part of the CARE team. The workshops will be held at a location selected by the school, likely on their campus.
  Interventions: Behavioral: Cultivating Awareness and Resilience in Education (CARE)

INTERVENTIONS:
Behavioral: Cultivating Awareness and Resilience in Education (CARE) — CARE provides teachers and staff with tools and resources to reduce stress, prevent burnout, enliven teaching, and help students thrive socially, emotionally, and academically. CARE blends instruction with experiential activities, reflection, and discussion.

SUMMARY:
This study looks at school employees' mental health, well-being, and effectiveness before and after completing a professional development workshop. The participants' schools are offering the Cultivating Awareness and Resilience in Education (CARE) professional development workshop to all teachers, staff, and administrators. CARE will be presented in three in-person training sessions over two to three months during the school year.

People who participate in CARE are asked to answer questions about their demographic information, mental health, well-being, and effectiveness before the workshop and two times after completing the workshop. This consent form provides the necessary information for people interested in answering these questions to make an informed decision. This consent form is not for the professional development workshop. Taking part in the workshop and questionnaires is optional.

This study is being conducted because teachers, school staff, and children's mental health has declined since the beginning of the COVID-19 pandemic. The investigators hope to use information collected in this study to tell schools, local public health officials, and state leaders how best to support teachers' mental health and well-being.

There are minimal risks associated with this study. The greatest risk of this study is loss of confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Adult participant, defined as an adult (18 years or older) employed by a school working with youth in kindergarten through 12th grade.
* Fluent in the English language

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily D'Agostino, DPH, MS, MEd, Principal Investigator — Duke University
Locations (1):
- Caldwell County Schools, Lenoir, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: School employees (teachers and staff) from two school districts in North Carolina, Caldwell County and Washington County, participated in this study.
Pre-assignment Details: Administrative and Non-Administrative Staff groups were combined due to low enrollment in those groups. Per protocol, "If the number of workshop participants for the administrative or non-administrative staff group is less than 10, then these participants will be grouped together."
Groups:
- Staff, Administrative and Non-Administrative: Schools will offer all administrative and non-administrative staff the professional development program called Cultivating Awareness and Resilience in Education (CARE) . CARE will be presented in three in-person training sessions over two to three months during the school year. Tools include mindful awareness practices and caring and emotion skills training. Each intervention workshop includes 30 to 35 participants and a facilitator, who is part of the CARE team. The workshops will be held at a location selected by the school, likely on their campus.
  Cultivating Awareness and Resilience in Education (CARE): CARE provides teachers and staff with tools and resources to reduce stress, prevent burnout, enliven teaching, and help students thrive socially, emotionally, and academically. CARE blends instruction with experiential activities, reflection, and discussion.
Period: Overall Study
Arm/Group | Teachers | Staff, Administrative and Non-Administrative
Started | 37 | 16
Completed | 37 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teachers | Staff, Administrative and Non-Administrative | Total
Number analyzed (Participants) | 37 | 16 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 16 | 53
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 7 | 3 | 10
  Gender: Female | 29 | 12 | 41
  Gender: Non-binary | 1 | 0 | 1
  Gender: Not reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Asian/Filipino | 1 | 0 | 1
  Race/Ethnicity: Black/African American | 6 | 4 | 10
  Race/Ethnicity: White/Caucasian | 29 | 12 | 41
  Race/Ethnicity: Not reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 16 | 53
Current grade level [Number; unit: participants] — This question permitted the selection of multiple responses.
  participants
    Elementary School | 17 | 8 | 25
    Middle School | 2 | 3 | 5
    High School | 18 | 7 | 25
Years in current role [Mean (Standard Deviation); unit: years] | 11.3 (6.73) | 6.2 (5.88) | 9.8 (6.85)
Years at current grade level [Mean (Standard Deviation); unit: years] | 9.9 (6.83) | 6.9 (6.88) | 9 (6.92)
Years at current school [Mean (Standard Deviation); unit: years] | 8 (6.38) | 5.1 (4.79) | 7.1 (6.05)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Self-effectiveness of Teachers After Completion of the CARE (Cultivating Awareness and Resilience in Education) Workshop Using the Teachers' Sense of Efficacy Scale (TSES)
Description: The TSES is used for rating teachers' efficacy in engaging students, providing instructional strategies, and managing classrooms. Total scores range from 1 to 9, with higher scores indicating a greater sense of efficacy. Scores are also calculated for three subscales measuring engagement, instruction and management.
Time Frame: Prior to intervention (baseline), 1 week post intervention, 2 months post intervention
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Teachers | Staff, Administrative and Non-Administrative
Number analyzed (Participants) | 37 | 16
score on a scale
  Pre-intervention to one week post-intervention | 0.91 [.047 to 1.36] | 1.04 [0.16 to 2.07]
  Pre-intervention to two months post-intervention | 0.74 [0.28 to 1.19] | 0.80 [-0.36 to 1.95]

2. Primary Outcome: Change in Efficacy in Student Engagement of Teachers After Completion of the CARE (Cultivating Awareness and Resilience in Education) Workshop Using the Teachers' Sense of Efficacy Scale (TSES)
Description: The TSES is used for rating teachers' efficacy in engaging students, providing instructional strategies, and managing classrooms. Student engagement scores range from 1 to 9, with higher scores indicating a greater sense of efficacy.
Time Frame: Prior to intervention (baseline), 1 week post intervention, 2 months post intervention
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Teachers | Staff, Administrative and Non-Administrative
Number analyzed (Participants) | 37 | 16
score on a scale
  Pre-intervention to one week post-intervention | 1.18 [0.63 to 1.73] | 1.27 [0.38 to 2.25]
  Pre-intervention to two months post-intervention | 1.00 [0.47 to 1.51] | 0.92 [-0.23 to 1.99]

3. Primary Outcome: Change in Efficacy in Instructional Strategies of Teachers After Completion of the CARE (Cultivating Awareness and Resilience in Education) Workshop Using the Teachers' Sense of Efficacy Scale (TSES)
Description: The TSES is used for rating teachers' efficacy in engaging students, providing instructional strategies, and managing classrooms. Instructional strategies scores range from 1 to 9, with higher scores indicating a greater sense of efficacy.
Time Frame: Prior to intervention (baseline), 1 week post intervention, 2 months post intervention
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Teachers | Staff, Administrative and Non-Administrative
Number analyzed (Participants) | 37 | 16
score on a scale
  Pre-intervention to one week post-intervention | 0.73 [0.29 to 1.17] | 1.23 [0.27 to 2.39]
  Pre-intervention to two months post-intervention | 0.54 [0.00 to 1.04] | 0.75 [-0.61 to 2.07]

4. Primary Outcome: Change in Efficacy in Classroom Management of Teachers After Completion of the CARE (Cultivating Awareness and Resilience in Education) Workshop Using the Teachers' Sense of Efficacy Scale (TSES)
Description: The TSES is used for rating teachers' efficacy in engaging students, providing instructional strategies, and managing classrooms. Classroom management scores range from 1 to 9, with higher scores indicating a greater sense of efficacy.
Time Frame: Prior to intervention (baseline), 1 week post intervention, 2 months post intervention
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Teachers | Staff, Administrative and Non-Administrative
Number analyzed (Participants) | 37 | 16
score on a scale
  Pre-intervention to one week post-intervention | 0.81 [0.33 to 1.31] | 0.63 [-0.33 to 1.70]
  Pre-intervention to two months post-intervention | 0.68 [0.18 to 1.17] | 0.73 [-0.35 to 1.87]

5. Primary Outcome: Change in Emotional Exhaustion (EE) After Completion of the CARE Workshop Using the Maslach Burnout Inventory (MBI)
Description: The Maslach Burnout Inventory - Educator Survey is used for assessing burnout by identifying how educators view their jobs and the individuals with who they work. Scores are calculated for the three subscales measuring emotional exhaustion (EE), depersonalization (DP), and personal accomplishment (PA). The EE subscale has a minimum score of 0 and maximum score of 54. A higher score on the EE subscale reflects a worse outcome, because it indicates that the participant is experiencing emotional exhaustion more frequently.
Time Frame: Prior to intervention (baseline), 1 week post intervention, 2 months post intervention
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Teachers | Staff, Administrative and Non-Administrative
Number analyzed (Participants) | 37 | 16
score on a scale
  Pre-intervention to one week post-intervention | -7.67 [-13.69 to -1.57] | -1.52 [-10.76 to 7.18]
  Pre-intervention to two months post-intervention | -8.46 [-14.18 to -2.34] | -1.59 [-12.37 to 8.89]

6. Primary Outcome: Change in Depersonalization (DP) After Completion of the CARE Workshop Using the Maslach Burnout Inventory (MBI)
Description: The Maslach Burnout Inventory - Educator Survey is used for assessing burnout by identifying how educators view their jobs and the individuals with who they work. Scores are calculated for the three subscales measuring emotional exhaustion (EE), depersonalization (DP), and personal accomplishment (PA). The DP subscale has a minimum score of 0 and maximum score of 30. A higher score on the DP subscale reflects a worse outcome, because it indicates that the participant depersonalizes others more frequently.
Time Frame: Prior to intervention (baseline), 1 week post intervention, 2 months post intervention
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Teachers | Staff, Administrative and Non-Administrative
Number analyzed (Participants) | 37 | 16
score on a scale
  Pre-intervention to one week post-intervention | -0.31 [-2.70 to 2.13] | 1.19 [-2.25 to 4.98]
  Pre-intervention to two months post-intervention | -0.11 [-2.65 to 2.54] | 1.19 [-3.25 to 6.53]

7. Primary Outcome: Change in Personal Accomplishment (PA) After Completion of the CARE Workshop Using the Maslach Burnout Inventory (MBI)
Description: The Maslach Burnout Inventory - Educator Survey is used for assessing burnout by identifying how educators view their jobs and the individuals with who they work. Scores are calculated for the three subscales measuring emotional exhaustion (EE), depersonalization (DP), and personal accomplishment (PA). The PA subscale has a minimum score of 0 and maximum score of 48. A higher score on the PA subscale reflects a better outcome, because it indicates that the participant recognizes personal accomplishments more frequently.
Time Frame: Prior to intervention (baseline), 1 week post intervention, 2 months post intervention
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Teachers | Staff, Administrative and Non-Administrative
Number analyzed (Participants) | 37 | 16
score on a scale
  Pre-intervention to one week post-intervention | 3.50 [0.49 to 6.63] | 4.48 [-1.17 to 11.16]
  Pre-intervention to two months post-intervention | 3.01 [0.03 to 5.91] | 1.77 [-5.47 to 9.20]

8. Primary Outcome: Change in Anxiety in Teachers After Completion of the CARE Workshop Using the Generalized Anxiety Disorder 7 (GAD-7) Scale.
Description: The GAD-7 measures generalized anxiety traits. Scores range from 0 to 21, with higher scores indicating the respondent experienced increased frequency in anxiety-related symptoms.
Time Frame: Prior to intervention (baseline), 1 week post intervention, 2 months post intervention
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Teachers | Staff, Administrative and Non-Administrative
Number analyzed (Participants) | 37 | 16
score on a scale
  Pre-intervention to one week post-intervention | -3.59 [-6.21 to -0.76] | 0.54 [-5.02 to 6.08]
  Pre-intervention to two months post-intervention | -3.27 [-5.83 to -0.71] | -1.42 [-6.66 to 3.82]

9. Primary Outcome: Change in Depression After Completion of the CARE Workshop Using the Patient Health Questionnaire 8 (PHQ-8) Scale
Description: The PHQ-8 scale is used to provide a brief report on depression symptoms. Scores range from 0 to 24, with higher scores indicating that the respondent experiences depression related symptoms at a higher frequency.
Time Frame: Prior to intervention (baseline), 1 week post intervention, 2 months post intervention
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Teachers | Staff, Administrative and Non-Administrative
Number analyzed (Participants) | 37 | 16
score on a scale
  Pre-intervention to one week post-intervention | -3.64 [-6.17 to -0.78] | 1.43 [-3.24 to 6.32]
  Pre-intervention to two months post-intervention | -3.19 [-5.73 to -0.63] | 0.23 [-4.78 to 5.56]

10. Primary Outcome: Change in Stress After Completion of the CARE Workshop Using the Perceived Stress Scale (PSS) Scale
Description: The PSS scale measures the perception of stress by examining the degree to which situations in one's life are assessed as stressful. The PSS scale has a minimum score of 0 and maximum score of 16. A higher score on the PSS scale reflects a worse outcome, because it indicates that the participant perceives stress more frequently in their life.
Time Frame: Prior to intervention (baseline), 1 week post intervention, 2 months post intervention
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Teachers | Staff, Administrative and Non-Administrative
Number analyzed (Participants) | 37 | 16
score on a scale
  Pre-intervention to one week post-intervention | -1.59 [-3.03 to -0.12] | 1.25 [-0.50 to 2.96]
  Pre-intervention to two months post-intervention | -0.68 [-2.22 to 0.85] | 1.16 [-1.51 to 3.74]

11. Other Pre Specified Outcome: Perceptions of Self-resiliency and Classroom Management After Completing the CARE Workshop Using the Cultivating Awareness and Resilience in Education (CARE) Professional Development (PD) Scale
Description: The CARE PD scale measures the participants' perceived changes in self-resiliency and classroom management after completing CARE. The CARE Professional Development Program scale has a min score of 1 and max score of 5: A score of 4 or 5 indicates an improvement in resiliency skills and classroom management; a score of 3 indicates no change in resiliency skills and classroom management; a score of 1 or 2 indicates a decline in resiliency skills and classroom management.
Time Frame: 1 week post intervention, 2 months post intervention
Population: Participants with data collected at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teachers | Staff, Administrative and Non-Administrative
Number analyzed (Participants) | 37 | 16
score on a scale
  1 week post intervention: number analyzed (Participants) | 27 | 14
  1 week post intervention | 3.99 (0.60) | 3.63 (0.68)
  2 months post intervention: number analyzed (Participants) | 29 | 11
  2 months post intervention | 3.72 (0.71) | 3.41 (0.86)

12. Other Pre Specified Outcome: Perceptions of Students' Behavior and Academic Performance After Completing the CARE Workshop Using the Result of Cultivating Awareness and Resilience in Education (CARE) Scale
Description: The Result of CARE scale measures participants' perceived changes in students' behavior and academic performance after completing CARE. The Result of CARE scale has a min score of 1 and max score of 5: A score of 4 or 5 indicates an improvement in student behavior and academic performance; a score of 3 indicates no change in student behavior and academic performance; a score of 1 or 2 indicates a decline in student behavior and academic performance.
Time Frame: 1 week post intervention, 2 months post intervention
Population: Participants with data collected at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teachers | Staff, Administrative and Non-Administrative
Number analyzed (Participants) | 37 | 16
score on a scale
  1 week post intervention: number analyzed (Participants) | 27 | 14
  1 week post intervention | 3.64 (0.54) | 3.29 (0.63)
  2 months post intervention: number analyzed (Participants) | 29 | 11
  2 months post intervention | 3.70 (0.51) | 3.55 (0.48)

ADVERSE EVENTS:
Time Frame: Adverse Events were not collected.
Description: Adverse Events were not collected.
Arm/Group | Teachers | Staff, Administrative and Non-Administrative
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/64/NCT05574764/Prot_SAP_001.pdf
  • Informed Consent Form (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/64/NCT05574764/ICF_000.pdf